CLINICAL TRIAL: NCT03442439
Title: Stamford Group Family Nurture Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Martha G. Welch, MD, Associate Professor of Psychiatry (in Pediatrics and Pathology and Cell Biology), Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AAAR5518
Record Dates: First submitted 2018-02-02; First posted 2018-02-22 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Behavior Problem; Developmental Delay; Emotional Disturbances; Family Conflict
Keywords: Family Nurture Intervention; Martha G. Welch MD; Randomized Controlled Trial; Preschool Intervention; Pre-school Intervention; Multiple Family Group Intervention; Emotional Connection; Co-regulation
MeSH Terms: conditions — Mental Disorders; Learning Disabilities; Affective Symptoms | interventions — Nutritional Status

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition and Play Intervention (NPI) (Active Comparator): Half of the mother-child dyads who are enrolled into the study will be randomly assigned to the Nutrition and Play Intervention group.
  Interventions: Behavioral: Nutrition and Play Intervention
- Family Nurture Intervention (FNI) (Experimental): Half of the mother-child dyads who are enrolled into the study will be randomly assigned to the Family Nurture Intervention group.
  Interventions: Behavioral: Family Nurture Intervention

INTERVENTIONS:
Behavioral: Nutrition and Play Intervention — Mothers and children in the Nutrition and Play group will play educational and nutrition-focused games.
  Other Names: NPI
  Arms: Nutrition and Play Intervention (NPI)
Behavioral: Family Nurture Intervention — The mother-child pair will be asked to talk and play with each other as they customarily do. If the child becomes restless and dysregulated the mother will be coached by the Nurture Specialist to bring the child back into a calm state though sustained physical contact; comfort touch, soothing words, and eye contact.
  Other Names: FNI
  Arms: Family Nurture Intervention (FNI)

SUMMARY:
The purpose of this current study is to investigate the efficacy of a group model of Family Nurture Intervention in ameliorating behavioral problems in preschool-aged children. The behavioral, neurobiological and clinical insights gained from this project may eventually lead to better treatment of emotional, behavioral, and developmental disorders. The investigator hypothesizes that the children who are treated with Family Nurture Intervention (FNI), which incorporates interactive touch with vocal soothing, and family practice in comforting, will show increased emotional connection and mother child co-regulation with better results in the outcome measures in the short term and long term.

DETAILED DESCRIPTION:
There are several early intervention programs that are available for children with emotional, behavioral and developmental disorders, ranging from behavioral treatment and sensory exposure therapy to pharmaceutical treatments. Although improvements in behavior have resulted from these interventions, they are limited in numerous ways. They are usually time-consuming, both for the child and the teacher or clinician providing the intervention. In order to see an effect of the intervention, most children must engage in the intervention procedure for several years. Moreover, the effects of most current intervention procedures are minimal to moderate. Pharmaceutical prescriptions are often accompanied by undesirable side effects that may modulate behavior, emotion, and physiological functions. The behavioral, neurobiological, and clinical insights gained from this project may eventually lead to better treatment of emotional, behavioral and developmental disorders.

ELIGIBILITY:
Inclusion Criteria:

* Child is a singleton
* Mother can speak, read and write in English or Spanish
* Child is between the ages of 2-4 1/2 years at date of enrollment
* Mother is 18 years of age or older at the time of consent
* Child resides with mother
* Child demonstrates developmental deficit as measured by the Strengths and Difficulties Questionnaire (13 or higher on behavioral questions or 4 or less on prosocial questions)
* Mother and child deemed "emotionally unconnected" using the Welch Emotional Connection Scale (WECS) to score their five minute Welch Lap Test video
* Mother is able to commit to study schedule

Exclusion Criteria:

* The child has severe congenital anomalies or chromosomal anomalies including Downs syndrome and Cerebral palsy
* Child has a motor disability
* Mother sees or hears things that other people do not seem to see or hear
* Mother has trouble distinguishing whether something is real or part of imagination or dreams
* Mother is currently taking antipsychotic medications
* Mother or child have any medical conditions that might prevent them from participating in block play, mother holding child, or child sitting on mother's lap
* Mother has any current drug and/or alcohol abuse
* Mother is more than 4 months pregnant
* Mother is currently involved with Department of Children and Families
* The child has a diagnosis of Autism

Ages: 24 Months to 54 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2018-11-25 (Actual); Study Completion 2018-11-25 (Actual)

PRIMARY OUTCOMES:
Welch Emotional Connection Scale (WECS) Score | 12 months
  This is designed to measure emotional connection. Children will be asked to sit on their mother's lap for five minutes. This interaction will be video taped, and will be behaviorally coded using the Welch Emotional Connection Scale (WECS) and using a paradigm evaluated in Noldus coding software.
  The Welch Emotional Connection Scale (WECS) construct is emotional connection between mother and child, which we hypothesize predicts optimal development. There are four items on the WECS: Mutual Attraction, Mutual Vocal Exchange, Mutual Facial Engagement, and Mutual Sensitivity/Reciprocity. Each item is rated on a scale from 1 to 3 in 0.25 increments with a score of 3 considered optimal. At or below 2.25 on any individual item, or a total score below 9 means that the mother-child pair is not emotionally connected. There is also a binary question to the rater asking if the pair is emotionally connected - yes or no. The mother and child are scored as a pair, not individually.

CONTACTS AND LOCATIONS:
Overall Officials: Martha G Welch, MD, Principal Investigator — Columbia University
Locations (1):
- Stamford Childrens Learning Center, Stamford, Connecticut, United States